CLINICAL TRIAL: NCT00436124
Title: A Randomized, Open Label Study to Evaluate the Effect of Tamiflu on Viral Shedding and on Serum and Cytoplasmic Inflammatory Cytokine Concentrations in Patients With Laboratory-confirmed Influenza
Brief Title: A Study of Tamiflu (Oseltamivir) Treatment in Laboratory-Confirmed Influenza.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: poor recruitment, no patients were enrolled
Sponsor: Hoffmann-La Roche (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML20910
Record Dates: First submitted 2007-02-15; First posted 2007-02-16 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Oseltamivir

INTERVENTIONS:
Drug: oseltamivir [Tamiflu]

SUMMARY:
This study will evaluate the efficacy and safety of Tamiflu in patients with clinically-diagnosed influenza occurring during an influenza outbreak within the community. Patients will be randomized to receive Tamiflu 75mg bid orally plus support therapy (NSAIDs and antibiotics) or support therapy alone. The anticipated time on study treatment is <3 months, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-64 years of age;
* ambulatory;
* influenza-like illness;
* positive rapid assay for detection of influenza antigen.

Exclusion Criteria:

* presentation >36h after onset of symptoms;
* influenza-like symptoms outside an outbreak based on local surveillance activities;
* influenza vaccination between November 2006 and January 2007;
* receipt of antiviral therapy, systemic steroids or immunosuppressants within 2 weeks prior to study day 1.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2007-01 (Actual); Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Viral shedding; serum and intracellular concentrations of inflammatory cytokines (INFgamma, TNFalpha, IL-6, IL-12).

SECONDARY OUTCOMES:
Efficacy: Duration of illness, health and functional status, extent and severity of symptoms, incidence of resistant viruses. Safety: AEs.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Genova, Italy